CLINICAL TRIAL: NCT06543628
Title: Tadalafil Combined With Low-Energy Pulsed Ultrasound (LIPUS) for the Treatment of Erectile Dysfunction: A Prospective, Randomized Controlled Clinical Trial
Brief Title: Evaluation of Tadalafil Combined With LIPUS for Treating Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0401
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-08

CONDITIONS: Erectile Dysfunction
Keywords: Tadalafil; LIPUS; Randomized Controlled Trial; protocol
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Separate the person responsible for randomization and assignment from the outcome assessor, ensure that the evaluator does not have access to information for the participant group, and assign a unique code to the participant, and the evaluator is only exposed to the code without knowing the specific intervention behind it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment group (Experimental): Participants will take tadalafil once daily at a dose of 5 mg for 6 months, in combination with LIPUS applied twice a week for 4 weeks, with the cycle repeated after a 4-week interval without treatment.
  Interventions: Drug: Tadalafil 5mg; Device: LIPUS (Low Intensity Pulsed Ultrasound)
- Control group (Active Comparator): Participants will take tadalafil once daily at a dose of 5 mg for 6 months.
  Interventions: Drug: Tadalafil 5mg

INTERVENTIONS:
Drug: Tadalafil 5mg — Participants will take tadalafil once daily at a dose of 5 mg for 6 months.
  Other Names: Cialis
Device: LIPUS (Low Intensity Pulsed Ultrasound) — Participants will receive LIPUS treatment applied twice a week for 4 weeks, with the cycle repeated after a 4-week interval without treatment.
  Arms: Treatment group

SUMMARY:
This study aims to evaluate the clinical efficacy and histological changes of tadalafil combined with low-intensity pulsed ultrasound (LIPUS) in patients with erectile dysfunction (ED) through a randomized controlled trial.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is defined as the persistent inability to achieve and maintain a sufficient erection for satisfactory sexual performance for more than six months. Low-intensity pulsed ultrasound (LIPUS), a non-invasive therapy, improves the pathological changes in the corpora cavernosa and penile hemodynamics by promoting the regeneration of connective tissue, blood vessels, and cavernous nerves, as well as reducing inflammation.

This study will recruit 114 patients diagnosed with ED and use simple random sampling to allocate them into a treatment group and a control group in a 1:1 ratio. The treatment group will receive daily 5mg tadalafil combined with LIPUS therapy twice a week for 4 weeks, followed by a 4-week interval without LIPUS treatment, and then repeat the treatment. The control group will receive only daily 5mg tadalafil.

Efficacy will be evaluated primarily through the minimal clinically important difference (MCID) of the International Index of Erectile Function-5 (IIEF-5) at each follow-up point, combined with Erectile Hardness Score (EHS), penile blood flow parameters, and elasticity values for comprehensive assessment.

This trial may provide additional clinical evidence for the efficacy, safety, and cost-effectiveness of tadalafil combined with LIPUS in treating ED patients. The inclusion of penile blood flow parameters and two-dimensional shear wave elastography will help establish a comprehensive evaluation system combining ED symptoms with histological assessment, providing new methods for efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 65 years old.
* An International Index of Erectile Function-5 (IIEF-5) score of 21 or less.
* First-time diagnosis of erectile dysfunction (ED) without prior treatment from traditional Chinese or Western medicine.
* A stable heterosexual relationship for at least 3 months.
* Agreement to attempt sexual intercourse at least four times every four weeks during the study period.
* Signing of an informed consent form.

Exclusion Criteria:

* Erectile dysfunction caused by spinal/neural injury or radical prostatectomy.
* History of priapism or penile anatomical abnormalities.
* Use of a penile prosthesis.
* Severe and poorly controlled psychological disorders.
* Untreated endocrine disorders, such as hypogonadism, hypothyroidism, or pituitary dysfunction.
* History of myocardial infarction, stroke, life-threatening arrhythmias, or potential cardiovascular risks during sexual activity within the six months prior to enrollment.
* Inability to complete the participant records required for the trial.
* Allergic constitution and multiple drug allergies.

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2024-08-11 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
MCID based on IIEF-5 | 0 months, 2 months, 4 months, 6 months
  The primary outcome measure is based on the Minimum Clinically Important Difference (MCID) derived from the International Index of Erectile Function-5 (IIEF-5) scores. The MCID will be determined by the changes in IIEF-5 scores at 0 months, 2 months, 4 months, and 6 months. The IIEF-5 scale ranges from a minimum of 5 to a maximum of 25, with higher scores indicating better erectile function.

SECONDARY OUTCOMES:
IIEF-5 Score | 0 months, 2 months, 4 months, 6 months
  The secondary outcome measure is the change in the International Index of Erectile Function-5 (IIEF-5) scores at 0 months, 2 months, 4 months, and 6 months. The scale is titled International Index of Erectile Function-5 (IIEF-5), with a minimum score of 5 and a maximum score of 25. The interpretation of the scores is that higher scores indicate better erectile function.
EHS | 0 months, 2 months, 4 months, 6 months
  The scale title is Erection Hardness Score (EHS), with a minimum value of 1 and a maximum value of 4. A higher score indicates better erection hardness. The changes in the EHS will be measured at 0 months, 2 months, 4 months, and 6 months.
PSV | 0 months, 6 months
  The change in Peak Systolic Velocity (PSV) measured by Doppler ultrasound at 0 months and 6 months.
EDV | 0 months, 6 months
  The change in End-Diastolic Velocity (EDV) measured by Doppler ultrasound at 0 months and 6 months.
YM value at the tip of the corpus cavernosum | 0 months, 6 months
  The change in Young's Modulus (YM) value measured by elastography at 0 months and 6 months.
YM value at the base of the corpus cavernosum | 0 months, 6 months
  The change in Young's Modulus (YM) value measured by elastography at 0 months and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Bodong Lv, MD, Study Chair — 2ndAffiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- The 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Q, Lv B, Yu H, Fu Y, Xu R, Liao Z, Zhang X, Fu Y, Huang W, Huang X. Evaluation of tadalafil in combination with Low-Intensity Pulsed Ultrasound (LIPUS) for erectile dysfunction: a protocol for a randomized controlled trial (SPIRIT Compliant). Trials. 2025 Nov 25;26(1):591. doi: 10.1186/s13063-025-09298-4. PMID 41291823